CLINICAL TRIAL: NCT02776735
Title: An Open-label, Sequential, Ascending, Repeated Dose-finding Study of Sarilumab, Administered With Subcutaneous (SC) Injection, in Children and Adolescents, Aged 2 to 17 Years, With Polyarticular-course Juvenile Idiopathic Arthritis (pcJIA) Followed by an Extension Phase
Brief Title: An Open-label, Ascending, Repeated Dose-finding Study of Sarilumab in Children and Adolescents With Polyarticular-course Juvenile Idiopathic Arthritis (pcJIA)
Acronym: SKYPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRI13925; U1111-1177-3487 (Registry Identifier: ICTRP); 2015-003999-79 (EudraCT Number)
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Sarilumab (Experimental): Participants received one of three ascending dose regimens of sarilumab by subcutaneous (SC) injection based on body weight. All the participants received the selected dose regimen once this was identified. Sarilumab was given during 12-week core treatment phase followed by an extension treatment phase (144 weeks for 73 participants enrolled in dose-finding and second portions and 84 weeks for approximately 29 participants enrolled in third portion)
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form:Solution Route of administration: Subcutaneous
  Other Names: SAR153191 (REGN88)

SUMMARY:
Primary Objective:

To describe the pharmacokinetic (PK) profile of sarilumab in participants aged 2-17 years with Polyarticular-course Juvenile Idiopathic Arthritis (pcJIA) in order to identify the dose and regimen for adequate treatment of this population

Secondary Objective:

To describe the pharmacodynamic (PD) profile, the efficacy and the long-term safety of sarilumab in participants with pcJIA.

DETAILED DESCRIPTION:
For 73 participants enrolled in the dose-finding and second portions, the total study duration per participant was up to 166 weeks that consists of a 4- week screening, a 12-week core treatment phase, a 144-week extension phase, and a 6-week post-treatment follow-up. For 29 participants enrolled in the third portion, the total study duration per participant was up to 106 weeks that consists of a 4- week screening, a 12-week core treatment phase, a 84-week extension phase, and a 6-week post-treatment follow-up.

ELIGIBILITY:
Inclusion criteria :

* Male and female participants aged ≥2 and ≤17 years (or country specified age requirement) at the time of the screening visit.
* Diagnosis of rheumatoid factor-negative or rheumatoid factor positive polyarticular Juvenile Idiopathic Arthritis (JIA) subtype or oligoarticular extended JIA subtype according to the International League of Associations for Rheumatology (ILAR) 2001 Juvenile Idiopathic Arthritis Classification Criteria with at least 5 active joints as per American College of Rheumatology (ACR) definition for "active arthritis" at Screening
* Participant with an inadequate response to current treatment and considered as a candidate for a biologic disease modifying antirheumatic drug (DMARD) as per investigator's judgment

Exclusion criteria:

* Body weight <10 kg or >60 kg for participants enrolled in the 3 ascending dose cohorts, then body weight <10 kg for participants subsequently enrolled at the selected dose-regimen.
* If nonsteroidal anti-inflammatory drugs (NSAIDs) [including cyclo oxygenase-2 inhibitors (COX-2)] taken, dose stable for <2 weeks prior to the baseline visit and/or dosing prescribed outside of approved label.
* If non-biologic DMARD taken, dose stable for <6 weeks prior to the baseline visit or at a dose exceeding the recommended dose as per local labeling.
* If oral glucocorticoid taken, dose exceeding equivalent prednisone dose 0.5 mg/kg/day (or 30 mg/day) within 2 weeks prior to baseline.
* Use of parenteral or intra-articular glucocorticoid injection within 4 weeks prior to baseline.
* Prior treatment with anti-interleukin 6 (IL-6) or IL-6 receptor (IL-6R) antagonist therapies, including but not limited to tocilizumab or sarilumab.
* Treatment with any biologic treatment for pcJIA within 5 half-lives prior to the first dose of sarilumab.
* Treatment with a Janus kinase inhibitor within 4 weeks prior to the first dose of sarilumab; and treatment with growth hormone within 4 weeks prior to the first dose of sarilumab (the required off treatment periods and procedures may vary according to local requirements).
* Treatment with any investigational biologic or non-biologic product within 8 weeks or 5 half-lives prior to baseline, whichever is longer.
* Lipid lowering drug stable for less than 6 weeks prior to screening.
* Exclusion related to tuberculosis (TB).
* Exclusion criteria related to past or current infection other than tuberculosis.
* Any live, attenuated vaccine within 4 weeks prior to the baseline visit, such as varicella-zoster, oral polio, rubella vaccines. Killed or inactive vaccine may be permitted based on the Investigator's judgment.
* Exclusion related to history of a systemic hypersensitivity reaction to any biologic drug and known hypersensitivity to any constituent of the product.
* Laboratory abnormalities at the screening visit (identified by the central laboratory).
* Pregnant or breast-feeding female adolescent participants.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- Children's Hospital Los Angeles Site Number : 8400416, Los Angeles, California, United States
- Argentina (2):
  - Investigational Site Number : 0320060, CABA, Buenos Aires
  - Investigational Site Number : 0320004, San Miguel de Tucumán
- Investigational Site Number : 1240112, Montreal, Quebec, Canada
- Investigational Site Number : 1520016, Concepción, Región del Biobío, Chile
- Investigational Site Number : 2030041, Brno, Czechia
- Investigational Site Number : 2460040, Helsinki, Finland
- Investigational Site Number : 2500040, Paris, France
- Germany (4):
  - Investigational Site Number : 2760064, Berlin
  - Investigational Site Number : 2760061, Bremen
  - Investigational Site Number : 2760062, Hamburg
  - Investigational Site Number : 2760060, Sankt Augustin
- Investigational Site Number : 3800052, Roma, Italy
- Mexico (2):
  - Investigational Site Number : 4840061, Guadalajara, Jalisco
  - Investigational Site Number : 4840060, Monterrey, Nuevo León
- Investigational Site Number : 5280020, Utrecht, Netherlands
- Poland (5):
  - Investigational Site Number : 6160074, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160073, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160070, Lublin, Lubusz Voivodeship
  - Investigational Site Number : 6160071, Lodz, Lódzkie
  - Investigational Site Number : 6160072, Sosnowiec, Silesian Voivodeship
- Russia (3):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430062, Moscow
  - Investigational Site Number : 6430063, Moscow
- Spain (4):
  - Investigational Site Number : 7240050, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240052, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240053, Madrid
  - Investigational Site Number : 7240051, Valencia
- United Kingdom (2):
  - Investigational Site Number : 8260031, London, London, City of
  - Investigational Site Number : 8260033, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Group A: >=30kg and <=60kg and Group B: <30kg and >=10kg. Portion 1 of study enrolled participants into 3 dosing regimens (Cohort 1, 2 and 3). Cohort 1: dose capped at 150mg q2w (Group A:2mg/kg q2w; Group B:2.5mg/kg q2w). Cohort 2: dose capped at 200mg q2w (Group A:3mg/kg q2w; Group B:4mg/kg q2w). Cohort 3: dose capped at 150mg qw (Group A:2mg/kg qw; Group B:2.5mg/kg qw). All 3 cohorts in Portion 1 received 12-week core treatment phase and eligible participants entered 144-week extension phase.
Pre-assignment Details: After dose-finding portion, 200mg q2w dose was selected for continuation in study. Portion 1 participants from Cohorts 1 and 3 who continued into extension phase switched to this dose after dose was selected. Participants enrolled into Portions 2 and 3 started on selected dose of 200mg q2w capped dose (Group A: 3 mg/kg q2w; Group B: 4 mg/kg q2w) for extension phase (144 weeks for Portion 2 and 84 weeks for Portion 3). A total of 102 participants were enrolled in the study.
Groups:
- Cohort 1: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kilograms (kg) and <= 60 kg received sarilumab 2 mg/kg subcutaneous (SC) injection once every other week (q2w) for 12 weeks in core treatment phase. Eligible participants continued to receive 2 mg/kg SC injection q2w until the selected dose was found and then switched to selected dose of 3 mg/kg SC injection q2w in extension phase (portion 1: up to 144 weeks in extension phase).
- Cohort 1: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 2.5 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants continued to receive 2.5 mg/kg SC injection q2w until the selected dose was found and then switched to selected dose of 4 mg/kg SC injection q2w in extension phase (portion 1: up to 144 weeks in extension phase).
- Cohort 2: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 3 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants continued to receive 3 mg/kg SC injection q2w in extension phase (portions 1 and 2: up to 144 weeks in extension phase and portion 3: up to 84 weeks in extension phase).
- Cohort 2: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 4 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants continued to receive 4 mg/kg SC injection q2w in extension phase (portions 1 and 2: up to 144 weeks in extension phase and portion 3: up to 84 weeks in extension phase).
- Cohort 3: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 2 mg/kg SC injection once every week (qw) for 12 weeks in core treatment phase. Eligible participants continued to receive 2 mg/kg SC injection qw until the selected dose was found and then switched to selected dose of 3 mg/kg SC injection qw in extension phase (portion 1: up to 144 weeks in extension phase).
- Cohort 3: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 2.5 mg/kg SC injection qw for 12 weeks in core treatment phase. Eligible participants continued to receive 2.5 mg/kg SC injection qw until the selected dose was found and then switched to selected dose of 4 mg/kg SC injection qw in extension phase (portion 1: up to 144 weeks in extension phase).
Period: Overall Study
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Started | 7 | 6 | 43 | 31 | 6 | 9
Treated | 7 | 6 | 42 | 31 | 6 | 9
Completed | 6 | 6 | 38 | 27 | 6 | 7
Not Completed | 1 | 0 | 5 | 4 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated population included participants who signed informed consent and received at least 1 dose of the study treatment.
Groups:
- Cohort 1: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 2 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants continued to receive 2 mg/kg SC injection q2w until the selected dose was found and then switched to selected dose of 3 mg/kg SC injection q2w in extension phase (portion 1: up to 144 weeks in extension phase).
- Cohort 3: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 2 mg/kg SC injection qw for 12 weeks in core treatment phase. Eligible participants continued to receive 2 mg/kg SC injection qw until the selected dose was found and then switched to selected dose of 3 mg/kg SC injection qw in extension phase (portion 1: up to 144 weeks in extension phase).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg | Total
Number analyzed (Participants) | 7 | 6 | 42 | 31 | 6 | 9 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (3.3) | 6.5 (3.2) | 12.6 (3.0) | 5.4 (3.1) | 13.7 (3.0) | 4.8 (2.4) | 9.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 35 | 23 | 3 | 6 | 77
  Male | 2 | 1 | 7 | 8 | 3 | 3 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 3 | 39 | 28 | 4 | 8 | 88
  Not Reported | 0 | 1 | 2 | 3 | 0 | 1 | 7
  Unknown | 1 | 2 | 0 | 0 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of Sarilumab at Week 12
Description: The Cmax was defined as maximum serum concentration. The values reported are mean and standard deviation.
Time Frame: Pre-dose on Days 1, 3, 5, 8, 12 and Weeks 2, 4, 8 and 12
Population: The Pharmacokinetic (PK) analysis set included all participants in the safety population with at least 1 post-dose, non-missing serum concentration value. Only participants with data collected are reported.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 3 | 5 | 38 | 25 | 6 | 5
milligram per liter (mg/L) | 7.57 (4.14) | 13.7 (2.52) | 22.0 (8.07) | 33.6 (7.16) | 32.0 (7.27) | 31.0 (7.98)

2. Primary Outcome: Area Under the Serum Concentration Versus Time Curve Using the Trapezoidal Method During a Dose Interval (AUC0-t) of Sarilumab at Week 12
Description: The AUC0-t was defined as area under the concentration in serum versus time curve calculated using the trapezoidal method during a dose interval (tau). The values reported are mean and standard deviation.
Time Frame: Pre-dose on Days 1, 3, 5, 8, 12 and Weeks 2, 4, 8 and 12
Population: The PK analysis set included all participants in the safety population with at least 1 post-dose, non-missing serum concentration value. Only participants with data collected are reported.
Measure: Mean (Standard Deviation); unit: day*mg/L
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 3 | 5 | 38 | 25 | 6 | 5
day*mg/L | 61.4 (25.2) | 106 (36.8) | 212 (77.2) | 318 (90.0) | 202 (55.0) | 192 (60.7)

3. Primary Outcome: Concentration Before Treatment Administration During Repeated Dosing (Ctrough) of Sarilumab at Week 12
Description: The Ctrough was defined as concentration observed before treatment administration during repeated dosing from baseline to Week 12. The values reported are mean and standard deviation.
Time Frame: Pre-dose on Days 1, 3, 5, 8, 12 and Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 3 | 5 | 38 | 25 | 6 | 5
mg/L | 1.30 (0.952) | 1.32 (1.27) | 5.76 (3.57) | 9.88 (5.42) | 22.2 (7.12) | 23.2 (8.28)

4. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in High-Sensitivity C-reactive Protein (Hs-CRP) at Week 12
Description: Serum concentrations of hs-CRP was determined to assess the Pharmacodynamic (PD) effects of sarilumab. The values reported are mean and standard deviation.
Time Frame: Baseline (Day 1) and Week 12
Population: All treated population included participants who signed informed consent and received at least 1 dose of the study treatment. Only participants analyzed at baseline and Week 12 are reported.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 6 | 6 | 9
mg/L | -1.00 (2.53) | -0.52 (3.64) | -5.71 (8.90) | -6.83 (11.74)

5. Secondary Outcome: Cohort 2: Change From Baseline in High-Sensitivity C-reactive Protein at Weeks 12, 24, 48, 96, and 156
Description: Serum concentrations of hs-CRP was determined to assess the PD effects of sarilumab. The values reported are mean and standard deviation.
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: All treated population included participants who signed informed consent and received at least 1 dose of the study treatment. Participants in Cohorts 1 and 3 only participated in portion 1 and then switched to Dose 2 after the dose is selected. Therefore, only Cohort 2 participants analyzed at baseline and specific time points are reported.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 40 | 29
mg/L
  Week 12 | -3.54 (33.57) | -20.66 (48.35)
  Week 24: number analyzed (Participants) | 37 | 29
  Week 24 | -8.54 (19.17) | -11.72 (23.54)
  Week 48: number analyzed (Participants) | 38 | 27
  Week 48 | -9.93 (21.60) | -12.57 (24.23)
  Week 96: number analyzed (Participants) | 36 | 23
  Week 96 | -9.39 (21.65) | -13.88 (25.96)
  Week 156: number analyzed (Participants) | 16 | 16
  Week 156 | -5.10 (14.68) | -12.30 (26.69)

6. Secondary Outcome: Change From Baseline in Interleukin-6 (IL-6) at Week 12
Description: Serum concentrations of IL-6 was determined to assess the PD effects of sarilumab. The values reported are mean and standard deviation.
Time Frame: Baseline (Day 1) and Week 12
Population: All treated population included participants who signed informed consent and received at least 1 dose of the study treatment. Only participants with data collected at Baseline and Week 12 are reported.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/L
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 4 | 4 | 30 | 20 | 6 | 5
nanogram (ng)/L | 1.27 (9.79) | 13.65 (18.20) | 43.71 (113.42) | 11.36 (35.81) | 66.21 (86.21) | 9.20 (26.50)

7. Secondary Outcome: Change From Baseline in Total Soluble Interleukin-6 Receptor (sIL-6R) at Week 12
Description: Serum concentrations of sIL-6R was determined to assess the PD effects of sarilumab. The values reported are mean and standard deviation.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 3 | 3 | 33 | 28 | 6 | 6
ng/mL | 40.09 (49.75) | 101.50 (129.59) | 316.77 (129.29) | 388.33 (185.82) | 535.76 (98.12) | 582.95 (149.52)

8. Secondary Outcome: Cohorts 1 and 3: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology (JIA ACR) 30 Response at Week 12
Description: JIA ACR30 response was defined as a participant with at least 3 out of the 6 JIA core set variables with >= 30% improvement from baseline with no more than 1 of the remaining variables worsened by >= 30%.
Time Frame: Week 12
Population: The efficacy analysis set included all participants who received at least 1 dose of sarilumab. Only participants analyzed at Week 12 are reported.
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
percentage of participants with response | 100 | 100 | 100 | 100

9. Secondary Outcome: Cohort 2: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 30 Response at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 8
Time Frame: Weeks 12, 24, 48, 96, and 156
Population: The efficacy analysis set included all participants who received at least 1 dose of sarilumab. Participants in Cohorts 1 and 3 only participated in portion 1 and then switched to Dose 2 after the dose is selected. Therefore, only Cohort 2 participants analyzed at baseline and specific time points are reported.
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
percentage of participants with response
  Week 12 | 100 | 100
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | 100 | 100
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | 100 | 100
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | 97.2 | 100
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | 94.1 | 100

10. Secondary Outcome: Cohorts 1 and 3: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 50 Response at Week 12
Description: JIA ACR50 response was defined as a participant with at least 3 out of the 6 JIA core set variables with >= 50% improvement from baseline with no more than 1 of the remaining variables worsened by >= 30%.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
percentage of participants with response | 80.0 | 100 | 100 | 100

11. Secondary Outcome: Cohort 2: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 50 Response at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 10
Time Frame: Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
percentage of participants with response
  Week 12 | 94.9 | 96.6
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | 100 | 100
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | 100 | 100
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | 97.2 | 100
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | 94.1 | 100

12. Secondary Outcome: Cohorts 1 and 3: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 70 Response at Week 12
Description: JIA ACR70 response was defined as a participant with at least 3 out of the 6 JIA core set variables with >= 70% improvement from baseline with no more than 1 of the remaining variables worsened by >= 30%.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
percentage of participants with response | 60.0 | 40.0 | 100 | 100

13. Secondary Outcome: Cohort 2: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 70 Response at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 12
Time Frame: Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
percentage of participants with response
  Week 12 | 74.4 | 89.7
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | 87.2 | 96.3
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | 89.5 | 100
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | 97.2 | 100
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | 94.1 | 100

14. Secondary Outcome: Cohorts 1 and 3: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 90 Response at Week 12
Description: JIA ACR90 response was defined as a participant with at least 3 out of the 6 JIA core set variables with >= 90% improvement from baseline with no more than 1 of the remaining variables worsened by >= 30%.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
percentage of participants with response | 60.0 | 20.0 | 66.7 | 60.0

15. Secondary Outcome: Cohort 2: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 90 Response at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 14
Time Frame: Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
percentage of participants with response
  Week 12 | 43.6 | 48.3
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | 64.1 | 74.1
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | 68.4 | 88.5
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | 80.6 | 95.8
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | 76.5 | 100

16. Secondary Outcome: Cohorts 1 and 3: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 100 Response at Week 12
Description: JIA ACR100 response was defined as a participant with at least 3 out of the 6 JIA core set variables with >= 100% improvement from baseline with no more than 1 of the remaining variables worsened by >= 30%.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
percentage of participants with response | 0 | 0 | 33.3 | 40.0

17. Secondary Outcome: Cohort 2: Percentage of Participants With Juvenile Idiopatic Arthritis American College of Rheumatology 100 Response at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 16
Time Frame: Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Number; unit: percentage of participants with response
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
percentage of participants with response
  Week 12 | 12.8 | 24.1
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | 23.1 | 48.1
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | 42.1 | 53.8
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | 47.2 | 70.8
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | 52.9 | 87.5

18. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Activity Joint Count-71, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using visual analog scale (VAS), Childhood Health Questionnaire Disability Index (CHAQ-DI) and hs-CRP. Activity joint count-71 was calculated as sum (joints with active arthritis)*(71/number of joints with assessment).
Time Frame: Baseline (Day 1) and Week 12
Population: The efficacy analysis set included all participants who received at least 1 dose of sarilumab. Only participants analyzed at baseline and Week 12 are reported.
Measure: Mean (Standard Error); unit: joint
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
joint | -14.40 (2.159) | -11.20 (2.871) | -16.50 (4.137) | -14.40 (5.573)

19. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Activity Joint Count-71, at Weeks 12, 24, 48, 96, and 156
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. Activity joint count-71 was calculated as sum (joints with active arthritis)*(71/number of joints with assessment).
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: joint
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
joint
  Week 12 | -15.15 (1.511) | -12.38 (1.519)
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | -16.66 (1.497) | -13.26 (1.575)
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | -17.24 (1.547) | -13.73 (1.618)
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | -16.47 (1.682) | -13.79 (1.751)
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | -18.65 (2.334) | -13.88 (2.495)

20. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Limited Motion Joint Count, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. Limited motion joint count was calculated as sum (joints with limited motion)*(67/number of joints with assessment).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: joint
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
joint | -7.80 (2.083) | -5.80 (2.267) | -7.83 (2.600) | -13.00 (4.219)

21. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Limited Motion Joint Count, at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 20
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: joint
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
joint
  Week 12 | -9.71 (1.249) | -9.21 (1.540)
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | -10.40 (1.330) | -10.63 (1.559)
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | -10.99 (1.498) | -10.73 (1.525)
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | -11.14 (1.661) | -10.42 (1.493)
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | -11.29 (2.203) | -11.81 (2.550)

22. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Childhood Health Assessment Questionnaire Disability Index, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. The CHAQ questionnaire consists of 30 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. Each domain is scored on a 4 point scale ranges from 0 to 3: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do). An additional response of "not applicable" is available to indicate activities the participant is unable to perform because he/she is too young. The CHAQ-DI total score is the sum of the domain scores divided by the number of domains that have a non-missing score. This overall score ranges from 0 (best) to 3 (worst). Higher scores indicate worse outcome.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
units on a scale | -0.80 (0.242) | -1.08 (0.239) | -0.42 (0.173) | -0.75 (0.213)

23. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Childhood Health Assessment Questionnaire Disability Index, at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 22
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
units on a scale
  Week 12 | -0.77 (0.092) | -0.74 (0.113)
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | -0.90 (0.096) | -0.95 (0.132)
  Week 48: number analyzed (Participants) | 38 | 27
  Week 48 | -0.88 (0.084) | -1.08 (0.119)
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | -0.92 (0.109) | -1.13 (0.136)
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | -1.07 (0.163) | -1.20 (0.169)

24. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, C-Reactive Protein, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. Serum concentrations of hs-CRP was determined to assess the PD effects of sarilumab.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
mg/L | -1.00 (1.130) | -1.67 (1.139) | -5.71 (3.633) | -2.54 (1.845)

25. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, C-Reactive Protein, at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 24
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
mg/L
  Week 12: number analyzed (Participants) | 39 | 27
  Week 12 | -3.84 (5.437) | -20.66 (9.304)
  Week 24: number analyzed (Participants) | 37 | 29
  Week 24 | -8.54 (3.151) | -11.72 (4.371)
  Week 48: number analyzed (Participants) | 38 | 27
  Week 48 | -9.93 (3.505) | -12.57 (4.664)
  Week 96: number analyzed (Participants) | 36 | 23
  Week 96 | -9.39 (3.608) | -13.88 (5.414)
  Week 156: number analyzed (Participants) | 16 | 16
  Week 156 | -5.10 (3.671) | -12.30 (6.672)

26. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Physician Global Assessment of Disease Activity, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. Physician global assessment of disease activity was assessed on an anchored 100 mm horizontal VAS score ranging from 0 to 10 where 0 is considered the best disease activity (no disease activity) and 10 the worst (most disease activity). Higher scores indicate worse outcome.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
units on a scale | -3.56 (0.969) | -6.30 (0.397) | -4.55 (0.509) | -5.68 (1.163)

27. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Physician Global Assessment of Disease Activity, at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 26
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
units on a scale
  Week 12 | -4.50 (0.248) | -4.09 (0.367)
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | -4.99 (0.237) | -5.01 (0.341)
  Week 48: number analyzed (Participants) | 38 | 26
  Week 48 | -5.27 (0.263) | -5.25 (0.321)
  Week 96: number analyzed (Participants) | 36 | 24
  Week 96 | -5.30 (0.306) | -5.35 (0.347)
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | -5.66 (0.396) | -5.73 (0.437)

28. Secondary Outcome: Cohorts 1 and 3: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Participant/Parent Assessment of Overall Well-Being, at Week 12
Description: The JIA ACR components included joints with active arthritis (0 to 71 joints), joints with limited motion (0 to 67 joints), physician global assessment of disease activity and participant/parent assessment of overall well-being using VAS, CHAQ-DI and hs-CRP. Participant/parent assessment of overall well-being was rated on an anchored 100 mm horizontal VAS score ranging from 0 to 10 where 0 is considered the best disease activity (no disease activity) and 10 the worst (most disease activity). Higher scores indicate worse outcome.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 5 | 5 | 6 | 5
units on a scale | -3.30 (1.014) | -3.16 (1.364) | -3.05 (0.992) | -5.00 (0.969)

29. Secondary Outcome: Cohort 2: Change From Baseline in Juvenile Idiopatic Arthritis American College of Rheumatology Component, Participant/Parent Assessment of Overall Well-Being, at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 28
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 39 | 29
units on a scale
  Week 12 | -3.73 (0.335) | -4.01 (0.435)
  Week 24: number analyzed (Participants) | 39 | 27
  Week 24 | -4.38 (0.313) | -4.39 (0.475)
  Week 48: number analyzed (Participants) | 38 | 27
  Week 48 | -4.21 (0.356) | -4.64 (0.510)
  Week 96: number analyzed (Participants) | 36 | 23
  Week 96 | -4.36 (0.387) | -5.09 (0.521)
  Week 156: number analyzed (Participants) | 17 | 16
  Week 156 | -4.19 (0.738) | -5.01 (0.636)

30. Secondary Outcome: Cohorts 1 and 3: Mean Change From Baseline in Juvenile Arthritis Disease Activity Score (JADAS-27) at Week 12
Description: The JADAS is used for assessment of disease activity, and it includes 4 measures: Physician global assessment of disease activity (VAS range: 0 to10; where 0= no activity and 10= maximum activity), parent/participant global assessment of well-being (VAS range: 0 to 10; where 0= no activity and10= maximum activity), count of joints with active disease (range: 0 to 27; where 0= no activity and 27= maximum activity), and index of inflammation determined by hs-CRP or ESR (normalized scale range: 0 to 10; where 0= no disease activity and 10= maximum disease activity). The JADAS total score is calculated as the simple sum of the scores of its 4 components. The total score ranges from 0 to 57 where 0= no disease activity and 57= maximum disease activity. Higher scores indicate higher disease activity. Clinical JADAS-27 is without CRP or ESR component and score ranges from 0 to 47 where 0= no disease activity and 47= maximum disease activity.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 18
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 7 | 6 | 6 | 9
units on a scale
  JADAS-27-ESR: Week 12: number analyzed (Participants) | 5 | 5 | 6 | 4
  JADAS-27-ESR: Week 12 | -15.4 (2.98) | -19.1 (3.05) | -20.0 (3.82) | -19.4 (6.01)
  JADAS-27-CRP: Week 12: number analyzed (Participants) | 5 | 5 | 6 | 5
  JADAS-27-CRP: Week 12 | -16.0 (2.78) | -18.1 (2.62) | -18.5 (3.42) | -21.1 (4.96)
  Clinical JADAS-27: Week 12: number analyzed (Participants) | 5 | 5 | 6 | 5
  Clinical JADAS-27: Week 12 | -16.1 (2.77) | -18.1 (2.62) | -18.3 (3.28) | -21.1 (4.96)

31. Secondary Outcome: Cohort 2: Mean Change From Baseline in Juvenile Arthritis Disease Activity Score at Weeks 12, 24, 48, 96, and 156
Description: as for outcome 30
Time Frame: Baseline (Day 1) and Weeks 12, 24, 48, 96, and 156
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg
Number analyzed (Participants) | 42 | 31
units on a scale
  JADAS-27-ESR: Week 12: number analyzed (Participants) | 37 | 29
  JADAS-27-ESR: Week 12 | -18.9 (1.46) | -16.9 (1.51)
  JADAS-27-ESR: Week 24: number analyzed (Participants) | 39 | 24
  JADAS-27-ESR: Week 24 | -21.9 (1.32) | -18.3 (1.72)
  JADAS-27-ESR: Week 48: number analyzed (Participants) | 38 | 26
  JADAS-27-ESR: Week 48 | -22.3 (1.45) | -19.4 (1.61)
  JADAS-27-ESR: Week 96: number analyzed (Participants) | 36 | 22
  JADAS-27-ESR: Week 96 | -22.4 (1.69) | -20.4 (1.84)
  JADAS-27-ESR: Week 156: number analyzed (Participants) | 16 | 14
  JADAS-27-ESR: Week 156 | -23.2 (2.06) | -20.6 (2.57)
  JADAS-27-CRP: Week 12: number analyzed (Participants) | 39 | 26
  JADAS-27-CRP: Week 12 | -18.2 (1.26) | -16.3 (1.42)
  JADAS-27-CRP: Week 24: number analyzed (Participants) | 37 | 27
  JADAS-27-CRP: Week 24 | -20.9 (1.20) | -18.8 (1.53)
  JADAS-27-CRP: Week 48: number analyzed (Participants) | 38 | 26
  JADAS-27-CRP: Week 48 | -21.6 (1.23) | -19.4 (1.58)
  JADAS-27-CRP: Week 96: number analyzed (Participants) | 35 | 21
  JADAS-27-CRP: Week 96 | -21.9 (1.58) | -20.1 (1.50)
  JADAS-27-CRP: Week 156: number analyzed (Participants) | 16 | 16
  JADAS-27-CRP: Week 156 | -21.8 (2.01) | -20.2 (2.24)
  Clinical JADAS-27: Week 12: number analyzed (Participants) | 39 | 29
  Clinical JADAS-27: Week 12 | -17.9 (1.19) | -16.0 (1.32)
  Clinical JADAS-27: Week 24: number analyzed (Participants) | 39 | 27
  Clinical JADAS-27: Week 24 | -20.5 (1.14) | -18.0 (1.46)
  Clinical JADAS-27: Week 48: number analyzed (Participants) | 38 | 26
  Clinical JADAS-27: Week 48 | -21.0 (1.22) | -18.8 (1.49)
  Clinical JADAS-27: Week 96: number analyzed (Participants) | 36 | 23
  Clinical JADAS-27: Week 96 | -21.2 (1.52) | -19.5 (1.60)
  Clinical JADAS-27: Week 156: number analyzed (Participants) | 17 | 16
  Clinical JADAS-27: Week 156 | -21.2 (1.85) | -19.3 (2.14)

32. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An adverse events (AEs) is any untoward medical occurrence in a participant or in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with the study treatment. An SAE is any untoward medical occurrence that at any dose results in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect or is an important medical event. TEAEs are defined as AEs that develop or worsen during the on-treatment period [that is, from the time of first dose of study treatment up to 6 weeks after the last administration of the study treatment].
Time Frame: From the first administration of study treatment (Day 1) up to end of treatment period, maximum of 156 weeks for portions 1 and 2 and 96 weeks for portion 3
Population: The Safety analysis set included all participants who received at least 1 dose or part of a dose of the study treatment, analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 7 | 6 | 42 | 31 | 6 | 9
Participants
  Any TEAE | 7 | 6 | 40 | 30 | 5 | 9
  Any treatment emergent SAE | 2 | 0 | 3 | 3 | 0 | 0

33. Secondary Outcome: Number of Participants With Local Site Reactions
Description: Participants were observed for at least 30 minutes after each study treatment administration either on site or at home and any local reactions were noted in the diary regardless of being clinically significant.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2: >= 30 kg and <= 60 kg | Cohort 2: < 30 kg and >= 10 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 3: < 30 kg and >= 10 kg
Number analyzed (Participants) | 7 | 6 | 42 | 31 | 6 | 9
Participants | 1 | 0 | 21 | 19 | 3 | 1

ADVERSE EVENTS:
Time Frame: From the first administration of study treatment (Day 1) up to end of study, maximum of 162 weeks for portions 1 and 2 and 102 weeks for portion 3.
Description: Analysis was performed on the safety analysis set.
Groups:
- Cohort 1: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 2 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants entered extension phase (up to 144 weeks) and continued to receive 2 mg/kg SC injection q2w until the selected dose 2 (3 mg/kg) was defined.
- Cohort 2 (From Baseline): >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 3 mg/kg SC injection q2w during the entire treatment period.
- Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 3 mg/kg SC injection q2w after switched from Dose/Cohort 1 to selected Dose 2.
- Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 3 mg/kg SC injection q2w after switched from Dose/Cohort 3 to selected Dose 2.
- Cohort 3: >= 30 kg and <= 60 kg: Participants with body weight >= 30 kg and <= 60 kg received sarilumab 2 mg/kg SC injection qw for 12 weeks in core treatment phase. Eligible participants entered extension phase (up to 144 weeks) and continued to receive 2 mg/kg SC injection q2w until the selected dose 2 (3 mg/kg) was defined.
- Cohort 1: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 2.5 mg/kg SC injection q2w for 12 weeks in core treatment phase. Eligible participants entered extension phase (up to 144 weeks) and continued to receive 2 mg/kg SC injection q2w until the selected dose 2 (3 mg/kg) was defined.
- Cohort 2 (From Baseline): < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 4 mg/kg SC injection q2w during the entire treatment period.
- Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 4 mg/kg SC injection q2w after switched from Dose/Cohort 1 to selected Dose 2.
- Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 4 mg/kg SC injection q2w after switched from Dose/Cohort 3 to selected Dose 2.
- Cohort 3: < 30 kg and >= 10 kg: Participants with body weight < 30 kg and >= 10 kg received sarilumab 2.5 mg/kg SC injection qw for 12 weeks in core treatment phase. Eligible participants entered extension phase (up to 144 weeks) and continued to receive 2 mg/kg SC injection q2w until the selected dose 2 (3 mg/kg) was defined.
Arm/Group | Cohort 1: >= 30 kg and <= 60 kg | Cohort 2 (From Baseline): >= 30 kg and <= 60 kg | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: >= 30 kg and <= 60 kg | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: >= 30 kg and <= 60 kg | Cohort 3: >= 30 kg and <= 60 kg | Cohort 1: < 30 kg and >= 10 kg | Cohort 2 (From Baseline): < 30 kg and >= 10 kg | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: < 30 kg and >= 10 kg | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: < 30 kg and >= 10 kg | Cohort 3: < 30 kg and >= 10 kg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/42 | 0/4 | 0/6 | 0/6 | 0/6 | 0/31 | 0/5 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/42 | 0/4 | 0/6 | 0/6 | 0/6 | 3/31 | 0/5 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 39/42 | 4/4 | 5/6 | 5/6 | 6/6 | 29/31 | 5/5 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: >= 30 kg and <= 60 kg (N=7) | Cohort 2 (From Baseline): >= 30 kg and <= 60 kg (N=42) | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: >= 30 kg and <= 60 kg (N=4) | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: >= 30 kg and <= 60 kg (N=6) | Cohort 3: >= 30 kg and <= 60 kg (N=6) | Cohort 1: < 30 kg and >= 10 kg (N=6) | Cohort 2 (From Baseline): < 30 kg and >= 10 kg (N=31) | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: < 30 kg and >= 10 kg (N=5) | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: < 30 kg and >= 10 kg (N=5) | Cohort 3: < 30 kg and >= 10 kg (N=9)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic Pseudocyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious Mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: >= 30 kg and <= 60 kg (N=7) | Cohort 2 (From Baseline): >= 30 kg and <= 60 kg (N=42) | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: >= 30 kg and <= 60 kg (N=4) | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: >= 30 kg and <= 60 kg (N=6) | Cohort 3: >= 30 kg and <= 60 kg (N=6) | Cohort 1: < 30 kg and >= 10 kg (N=6) | Cohort 2 (From Baseline): < 30 kg and >= 10 kg (N=31) | Cohort 1 Portion 1, Post Dose-adjustment From Dose 1: < 30 kg and >= 10 kg (N=5) | Cohort 3 Portion 1, Post Dose-adjustment From Dose 3: < 30 kg and >= 10 kg (N=5) | Cohort 3: < 30 kg and >= 10 kg (N=9)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 10 (23) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 15 (78) | 2 (2) | 0 (0) | 6 (9)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental Discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (6) | 0 (0) | 1 (1) | 2 (2)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulpless Tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 1 (1)
Administration Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Erythema (General disorders) | 1 (1) | 4 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Injection Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Injection Site Urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy To Arthropod Bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 2 (5)
Covid-19 (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eczema Impetiginous (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 9 (11) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Groin Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious Mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum Contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 11 (21) | 0 (0) | 4 (6) | 3 (5) | 1 (1) | 17 (38) | 0 (0) | 3 (5) | 3 (6)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (11) | 1 (2)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Otitis Media Acute (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Pharyngitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 1 (1) | 2 (5) | 3 (3)
Scarlet Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (10) | 6 (10) | 3 (5) | 1 (2) | 2 (2) | 2 (2) | 3 (6) | 0 (0) | 1 (1) | 2 (3)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Systolic Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eosinophil Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Mean Cell Volume Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Monocyte Count Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Monocyte Count Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (2)
Affective Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (9) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis Alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urticaria Chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02776735/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02776735/SAP_001.pdf